CLINICAL TRIAL: NCT01471119
Title: Usefulness and Safety of Sublingual Dermatophagoides Farinae Drops in Patients With Atopic Dermatitis:A Randomized,Double-blind,Placebo-controlled Study.
Brief Title: Sublingual Immunotherapy in Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Wolwo Bio-pharmaceutical Co. LTD. (Unknown); Huashan Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Peking University Third Hospital (Other); Tongji Hospital (Other); First Affiliated Hospital of Suzhou Medical College (Other)
Responsible Party: Principal Investigator, Min Zheng, Director of dermatology department,Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WOLWO-CT-A1.0
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2015-08

CONDITIONS: Atopic Dermatitis
Keywords: sublingual immunotherapy; atopic dermatitis; Dermatophagoides Farinae Drops
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dermatophagoides Farinae Drops Group 1 (Experimental): Dermatophagoides Farinae Drops Group 1 is the group with maintenance dose of 2 drops of grade 5 Dermatophagoides Farinae and 1 drop of placebo.
  Interventions: Biological: Dermatophagoides Farinae Drops Group 1
- Dermatophagoides Farinae Drops Group 2 (Experimental): Dermatophagoides Farinae Drops Group 2 is the group with maintenance dose of one drop of grade 5 Dermatophagoides Farinae and 2 drops of placebo.
  Interventions: Biological: Dermatophagoides Farinae Drops Group 2
- Dermatophagoides Farinae Drops Group 3 (Experimental): Dermatophagoides Farinae Drops Group 3 is the group with maintenance dose of 3 drops of grade 4 Dermatophagoides Farinae.
  Interventions: Biological: Dermatophagoides Farinae Drops Group 3
- Placebo (Experimental): Placebo Group is the group with maintenance dose of 3 drops of placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Dermatophagoides Farinae Drops Group 1 — Dermatophagoides Farinae Drops Group 1 is the group with maintenance dose of 2 drops of grade 5 Dermatophagoides Farinae and 1 drop of placebo.
  Arms: Dermatophagoides Farinae Drops Group 1
Biological: Dermatophagoides Farinae Drops Group 2 — Dermatophagoides Farinae Drops Group 2 is the group with maintenance dose of one drop of grade 5 Dermatophagoides Farinae and 2 drop of placebo.
  Arms: Dermatophagoides Farinae Drops Group 2
Biological: Dermatophagoides Farinae Drops Group 3 — Dermatophagoides Farinae Drops Group 3 is the group with maintenance dose of 3 drops of grade 4 Dermatophagoides Farinae.
  Arms: Dermatophagoides Farinae Drops Group 3
Biological: Placebo — Placebo Group is the group with maintenance dose of 3 drops of placebo.
  Arms: Placebo

SUMMARY:
To assess the effect and safety of sublingual Dermatophagoides Farinae Drops in adult patients with atopic dermatitis and allergic sensitization to house dust mites.240 adults age 18 to 60 years with atopic dermatitis(Objective Scoring Atopic Dermatitis, Objective SCORAD from 10 to 40) are going to be enrolled in a randomized,double-blind,placebo-controlled study.Sublingual Dermatophagoides Farinae Drops or placebo is given for 9 months in addition to standard therapy.SCORAD,average anesis interval,rescue medicine and DLQI will be recorded.

DETAILED DESCRIPTION:
SCORAD is composed of skin rash area,severity and subjective symptom including pruritus and sleeping quality.Skin rash area and severity score are objective SCORAD(range from 0 to 83).Subjective SCORAD range from 0 to 20 and total SCORAD range from 0 to 103.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex ,aged from 18 to 60 years. Diagnosed of atopic dermatitis.
* Mild to moderate AD ( [SCORAD] 1O-40)
* The results of skin prick tests with dermatophagoides farinae allergen extracts preparation is positive(≥2+)
* Written informed consent by the subject or legal guardian.
* Female patients of child-bearing potential must be negative pregnant test on screening and use an appropriate method of contraception.

Exclusion Criteria:

* Dust mites are not the primary allergens.
* Pregnant, breastfeeding women or women planned to pregnant within 1 year.
* Have concurrent skin disease that it could interfere with the study evaluation.
* Were treated with antihistamines or topical therapy within 7 days of randomization.
* Have received systemic corticosteroids,leukotriene receptor antagonists or immunosuppressants within 4 weeks of randomization.
* Have received phototherapy (e.g. UVA, UVB) within 4 weeks of randomization.
* Have a history of immune suppressed diseases(malignant tumor or infection of HIV), autoimmune disease or tuberculosis.
* Patients with impaired liver function (aspartate aminotransferase and/ or alanine aminotransferase levels 1.5 times the upper limit of normal), impaired renal function(serum creatinine>normal value) or other severe diseases.
* Bronchial asthma patients who need treatments with corticosteroids and or β agonists(including injection, oral administration or inhalation) regularly.
* Patients who need to take β-blockers during research.
* Have received investigational drugs within 3 months prior to randomization or planned use of other investigational drugs during participation in this study.
* Have received immunotherapy with dust mite preparation within 3 years prior to randomization.
* Patients with severe mental disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 239 (Actual)
Dates: Start 2011-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
average anesis interval | baseline and 36 week
  The average duration of last 3 whole anesis interval.
Rescue medication consumption | 36 week
  The total sum of rescue medication consumption will be recorded.
SCORAD | baseline and 36 week
  Change of SCORAD will be assessed.

SECONDARY OUTCOMES:
DLQI | baseline and 36 week
  Change of Dermatology Life Quality Index will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Min Zheng, Doctor, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital,School of Medicine,Zhejiang University., Hangzhou, Zhejiang, China